CLINICAL TRIAL: NCT07352085
Title: Exoskeleton-assisted Neurorehabilitation: Current Perspectives and Future Directions - A Pilot Study
Brief Title: Exoskeleton-assisted Neurorehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, Head of Department, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IKEB2023/10
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Spinal Cord Injuries (Complete and Incomplete); Cerebellar Ataxia; Spastic Paraplegia
Keywords: Spinal cord injury; Ataxia; Stroke; Spastic paraplegia; Altered gait pattern; Eksobionics; Robotic therapy
MeSH Terms: conditions — Stroke; Spinal Cord Injuries; Cerebellar Ataxia; Paraplegia; Ataxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ekso Group (Active Comparator): Improving gait with the help of the Eksobionics EksoNR device
  Interventions: Device: Gait training with exoskeleton

INTERVENTIONS:
Device: Gait training with exoskeleton — EksoNR is a wearable, battery-powered bionic exoskeleton that enables individuals with neurological or muscular injuries, lower limb weakness, paralysis, or gait disorders to stand and walk on flat surfaces. The hip and knee joints are powered by motors, and all movements are performed either by the patient's specific movements or by using an external controller. The robot's functions can be adjusted to determine the level of assistance the device provides to the patient.

SUMMARY:
* Objective assesment of the feasibility of integrating the Ekso Bionics - Ekso NR device into outpatient care
* Objective assesment of quality of life, functionality and clinical symptomps of patients with stroke, cerebellar ataxia, spinal cord injury, and spastic paraparesis
* Comparison of measured data and follow-up of changes in relation to themselves and each other
* Analyzing the effects of the exoskeleton among the patients
* Assessing the safety, possible side effects and tolerability of the EksoNR

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of spinal cord injury (at or below the C4 level)
* having cerebellar ataxia diagnosis
* confirmed spastic paraparesis
* ischemic stroke

Exclusion Criteria:

* height below 150 cm or above 190 cm
* body weight exceeded 100 kg
* multiple strokes in medical history
* systolic blood pressure less than 120 or higher than 160 mmHg
* orthostatic hypotension
* arotid artery stenosis
* severe heart disease
* hemophilia
* traumatic brain injury
* seizure disorder
* untreated diabetes
* abnormal electroencephalography
* abnormal blood panel
* use of sedatives
* irregular medication use
* severe aphasia (Western Aphasia Battery ≤ 25)
* severe visual or hearing impairment
* severe sensory dysfunction
* severe orthopedic problems
* alcoholism
* drug use
* smoking after diagnosis of stroke
* unable to walk at least 10 m with or without assistance in 6 minutes
* BBS score ≤ 32
* BI score ≤ 70
* current participation in individual or group exercise program outside of standard physical therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) | 4 weeks
  Functional autonomy, scaling 18-126 points. The lower the score, the less self-sufficient the patient is.
Barthel Index (BI) | 4 weeks
  Everyday activities, scaling 0-100 points. The higher the score, the better the self-sufficiency.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) | 4 weeks
  Measures functional mobility and fall risk, scaling 0-180 seconds. The less time, the lower the risk of falling.
Berg Balance Scale (BBS) | 4 weeks
  Measures balance, scaling 0-56 points, with lower scores suggesting good balance/indipandance.
Tinetti | 4 weeks
  Balance and walking, scaling 0-28 points, with lower scores indicating higher fall risk.
Walking Index for Spinal Cord Injury II. (WISCI II.) | 4 weeks
  21 - level ordinal scale scoring walking ability after SCI, from total depenence (0) to independent walking (20).
6 minute walk test (6MWT) | 4 weeks
  Functional exercise capacity, scaling 0-800 meters. The more meters a patient achieves, the better their cardiopulmonary function.
EG-5D-5L | 4 weeks
  Health-related quality of life, having 5 dimensions and 5 levels, plus a Visual Analogue Scale (EQ-VAS)
WHO Quality of Life (WHOQOL) | 4 weeks
  Measuring quality of life, scoring involves rating items on a 1-5 Likert scale, then tranforming these raw scores into a 0-100 scale for four main domains (Physical Health, Psychological, Social Relationships, Environment). The higher the score, the better the quality of life is.

CONTACTS AND LOCATIONS:
Overall Officials: József Dr. habil. Tollár, Principal Investigator — Somogy County Kaposi Mór Teaching Hospital
Locations (1):
- Somogy County Kaposi Mór Teaching Hospital, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No